CLINICAL TRIAL: NCT04731194
Title: Promoting the Adoption of Local Government Policy on the Reimbursement of Chronic Disease Medicines (PAPMed): a Field-based Cluster-Randomized Controlled Trial in Rural Nantong, China
Brief Title: Promoting Medication Reimbursement Policy (PAPMed)
Acronym: PAPMed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duke Kunshan University (Other)
Collaborators: Duke University (Other); Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020DUKE0002
Record Dates: First submitted 2021-01-14; First posted 2021-01-29 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Chronic Illness
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- performance-based financial incentive program (Experimental): Village doctors in villages of the intervention group will promote policy awareness, support registration, follow-up patients, and receive financial incentives based on their performance.
  Interventions: Behavioral: Performance-based financial incentive program
- current situation (No Intervention): Village doctors in villages of the control group will not be contacted. The control group would serve as a natural baseline and do not receive any intervention.

INTERVENTIONS:
Behavioral: Performance-based financial incentive program — 1. Enhance policy awareness through verbal communication with patients, distributing picture-rich fliers to patients, and putting up large posters in public places of the villages.
  2. Support patients' registration in the reimbursement system
  3. Follow-up patients after the first, third, and sixth months after the start of the study, measuring blood pressure and blood glucose level. Encourage patients to purchase medications from public institutions and to take their medications on time.
  4. Receive financial incentives based on performance in the amount of 3 RMB per patient enrolled (first month) and 5 RMB per patient (at third and sixth month) buying medications with reimbursement from the policy.
  Arms: performance-based financial incentive program

SUMMARY:
Rationale: Chronic non-communicable diseases (NCDs) have become the leading cause of morbidity and mortality in China. Rural NCDs patients are more likely to suffer from poverty. Nantong city has established a reimbursement plan covering 50% of hypertension and diabetes medication costs, however, various barriers prevent patients from taking advantage of this policy. Objectives: To evaluate the effectiveness of the intervention on saving medical costs and promoting health in rural populations. Study design: a cluster-randomized controlled trial. Study population: village doctors and health insurance officials at township hospitals are implementors of the intervention. Patients in the basic public health service system are the target populations of the intervention. Randomization: 31 villages are included in the study. 1 village is randomly dropped, and the rest of the villages will be randomly assigned to the intervention and control group stratified by township with an allocation ratio of 1:1. Intervention and follow-up: village doctors will promote policy awareness and support patients registration. They will follow-up patients on the 1st, 3rd, and 6th month and receive financial incentives based on their performance of supporting patients registration and encouraging patients to buy medications in designated medical institutions to be reimbursed. Control: The control group would serve as a natural baseline and do not receive any intervention. Outcomes: Patients' registration rate, medical costs saved, medication compliance rate, and improvements on health indicators will be evaluated based on real-world medical examination, prescription, and insurance data. Sample size: an estimated sample of 5000 patients from 30 clusters will be registered in the policy.

DETAILED DESCRIPTION:
Rationale: Chronic non-communicable diseases (NCDs) have become the leading cause of morbidity and mortality in China. Rural NCDs patients are more likely to suffer from poverty. Nantong city has established a reimbursement plan covering 50% of hypertension and diabetes medication costs, however, various barriers prevent patients from taking advantage of this policy. Objectives: To evaluate the effectiveness of the intervention on saving medical costs and promoting health in rural populations. Study design: a cluster-randomized controlled trial. Study population: village doctors and health insurance officials at township hospitals are implementors of the intervention. Patients in the basic public health service system are the target populations of the intervention. Randomization: 31 villages are included in the study. 1 village is randomly dropped, and the rest of the villages will be randomly assigned to the intervention and control group stratified by township with an allocation ratio of 1:1. Intervention and follow-up: village doctors will promote policy awareness and support patients registration. They will follow-up patients on the 1st, 3rd, and 6th month and receive financial incentives based on their performance of supporting patients registration and encouraging patients to buy medications in designated medical institutions to be reimbursed. Control: The control group would serve as a natural baseline and do not receive any intervention. Outcomes: Patients' registration rate, medical costs saved, medication compliance rate, and improvements on health indicators will be evaluated based on real-world medical examination, prescription, and insurance data. Sample size: an estimated sample of 5000 patients from 30 clusters will be registered in the policy.

ELIGIBILITY:
Inclusion criteria:

To be eligible to register in the medication reimbursement policy, patients need to be:

1. Living in the service areas of the village clinics
2. Officially diagnosed with hypertension and/or diabetes in a township level hospital or above
3. Registered as a hypertensive and/or diabetic patient in the public health service system

Exclusion criteria:

Not part of the New Cooperative Medical Scheme (NCMS) for rural residents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Registration Rate | 6 months
  The percentage of patients registered to the policy in the health insurance system

SECONDARY OUTCOMES:
Registration number | 6 months
  The number of all registered patients in the village served by the village clinic
Medical costs saved | 6 months
  The amount of money saved on outpatient expenses, hospital expenses, personal out-of-pocket expenses, and medical insurance reimbursement expenses
Doctor visiting frequency | 6 months
  Rate and visiting frequency of registered patients seeing doctors in designated hospitals
Medication compliance rate | 6 months
  Prescription frequency and doses, medication purchasing rate among registered patients, times of reimbursement during intervention and follow-up period among registered patients, insulin usage rate among registered diabetic patients
Blood pressure | 6 months
  Average systolic and diastolic blood pressure level among all rural hypertensive patients
Blood glucose | 6 months
  Average blood glucose level among rural diabetic patients
Blood lipids | 6 months
  Average blood lipids level among rural hypertensive and diabetic patients

CONTACTS AND LOCATIONS:
Locations (1):
- Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He Z, Cao X, Zhao D, Tang Z, Zhao J, Beasley M, Renne A, Liu L, Zhu S, Gao Y, Yan LL. Promoting the adoption of local governmental policy on the reimbursement of chronic disease medicines (PAPMed): study protocol of a field-based cluster randomized trial in rural Nantong, China. Trials. 2022 Sep 15;23(1):785. doi: 10.1186/s13063-022-06710-1. PMID 36109757